CLINICAL TRIAL: NCT02115997
Title: A Study Evaluating the Safety and Efficacy of Rituximab in Combination With Glucocorticoids in Participants With Wegener's Granulomatosis or Microscopic Polyangitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28550
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Wegener's Granulomatosis or Microscopic Polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — Methylprednisolone; Prednisone; Rituximab

ARMS (1):
- Rituximab (Experimental): Participants will receive IV infusion of rituximab once weekly from Week 1 to 4. Participants will also receive one pulse of methylprednisolone, followed by a tapering dose of oral prednisolone at the discretion of the investigator. Methylprednisolone may be repeated up to total of 3 pulses at the discretion of the investigator.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone; Drug: Rituximab

INTERVENTIONS:
Drug: Methylprednisolone — Methyprednisolone will be administered 1 to 3 pulses at a dose of 1000 milligram (mg) IV at the discretion of the investigator.
Drug: Prednisone — Prednisone will be administered orally at tapered dose (start at 1 milligrams per kilogram per day [mg/kg/day]) at the discretion of investigator given daily until participants are off the drug.
Drug: Rituximab — Rituximab will be administered at 375 milligrams per meter square (mg/m^2) of body surface area given by IV infusion once weekly from Week 1 to 4.
  Other Names: Ristova

SUMMARY:
This is a perspective, Phase IV, multi-center, single arm, open-label, interventional study in adult participants with Wegener's granulomatosis (granulomatosis with polyangiitis [GPA]) or microscopic polyangiitis. Participants will be treated with rituximab (Ristova) and glucocorticoids. Rituximab will be administered by intravenous (IV) infusion at a dose of 375 milligrams per meter square (mg/m^2) body surface area once weekly during Weeks 1 to 4. Participants will also receive one or three pulses of methylprednisolone (1000 milligram [mg] each), followed by a tapering dose of oral prednisolone (start dose of 1 mg per kilogram per day). The dose of oral prednisone will be reduced as per evaluation by the investigator till the participant is completely off the drug. The participants will be followed up for duration of 6 months from the date of starting rituximab therapy with three follow-up visits at Days 52, 112 and 172. All adverse events occurring during this period will be captured.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-nursing female
* Diagnosed with Wegener's granulomatosis or Microscopic polyangiitis according to the definitions of the Chapel Hill Consensus Conference
* Participants with either newly diagnosed or relapsing disease
* Participants must have active disease as per the BVAS/WG greater than equal to (>/=) 3 that would normally require treatment with cyclophosphamide (CYC)
* Participants willing to practice medically acceptable contraception during and 1 year after the completion of rituximab therapy
* Participants must have severe disease i.e. one or more of the major BVAS/WG items depicting severity or disease severe enough to require treatment with CYC.
* Participants must be positive for either proteinase 3-antineutrophil cytoplasmic antibodies (PR3-ANCA) or myeloperoxidase-antineutrophil cytoplasmic antibodies (MPO-ANCA) at the screening

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Participants in a severely immunocompromised state
* Participants with severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Participants having active severe infection or history of recurrent bacterial, viral, fungal, mycobacterial or other infections
* Participants who had a live vaccine fewer than 4 weeks before first dose of rituximab
* Any other condition which puts the participant to undue risk for rituximab therapy as per local prescribing information or Investigator's judgment
* Participants with any previous treatment with rituximab
* Participants with any previous treatment with alemtuzumab
* Participants who have had treatment with infliximab within the previous 3 months
* Participants who have had treatment with adalimumab within the previous 2 months
* Participants who have had treatment with etanercept within the previous month
* Participants with any other investigational medication within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events and Serious Adverse Events | Baseline up to 6 months
Percentage of Participants Who Achieved a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) Score of 0 and Successfully Completed Prednisone Taper at 6 Months | 6 months

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved a BVAS/WG Score of 0 During Treatment With Prednisone at a Dose of Less Than (<) 10 mg/day | 6 months
Percentage of Participants With Refractory Antineutrophil Cytoplasmic Antibodies-Associated Vasculitis (AAV) Who Achieved BVAS/WG Score of 0 and Successfully Completed Prednisone Taper at 6 Months | 6 months
Percentage of Participants Who Achieved and Maintained Partial Remission (Defined as Having a BVAS/WG of 1 or 2) | 6 months
Number of Severe Flares | At Months 2, 4, 6
Number of Limited Flares | At Months 2, 4, 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- India (10):
  - Yashoda Hospital, Hyderabad, Andhra Pradesh
  - MULJIBHAI PATEL UROLOGICAL HOSPITAL; Nephrology, Gujarat, Gujarat
  - Medanta-The Medicity, Gurgaon, Haryana
  - Fortis Memorial Research Instititute, Gurgaon, Haryana
  - Apollo BGS Hospitals, Mysuru, Karnataka
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute; Department of Rheumatologz, Mumbai, Maharashtra
  - St. John's Medical College Hospital; Rheumatology, Bangalore
  - Chanre Rheumatology and Immunology Center and Research, Bangalore
  - Jasleen Hospital, Nagpur
  - Fortis Hospital, Noida